CLINICAL TRIAL: NCT03990025
Title: A Prospective Randomized Study of Linked Color Imaging and Conventional White Light Imaging in Gastroscopy for the Detection of Gastric Cancer Precursors
Brief Title: Linked Color Imaging vs White Light Imaging for Detection of Gastric Cancer Precursors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Changi General Hospital (Other)
Collaborators: Singapore General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Diagnostic
Other Study IDs: 2018/2895
Record Dates: First submitted 2019-03-27; First posted 2019-06-18 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2020-01

CONDITIONS: Early Gastric Cancer; Barrett Esophagus
MeSH Terms: conditions — Stomach Neoplasms; Barrett Esophagus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Linked Color Imaging - White Light Imaging (Other): Participant undergoes gastroscopy via Linked Color Imaging first, then followed by White Light Imaging
  Interventions: Diagnostic Test: Linked Color Imaging; Diagnostic Test: White Light Imaging
- White Light Imaging - Linked Color Imaging (Other): Participant undergoes gastroscopy via White Light Imaging first, then followed by Linked Color Imaging
  Interventions: Diagnostic Test: Linked Color Imaging; Diagnostic Test: White Light Imaging

INTERVENTIONS:
Diagnostic Test: Linked Color Imaging — Linked Color Imaging (LCI) is a form of image enhanced endoscopy that uses a laser endoscopic system that acquires images by simultaneously using narrow-band wavelength light and white light in an appropriate balance. This enhances slight color differences in the red region of the mucosa.
Diagnostic Test: White Light Imaging — White Light Imaging (WLI) uses conventional white light that encompasses all bandwidths of light to illuminate areas of interest to obtain endoscopic images.

SUMMARY:
This study aims to examine the use of Linked Color Imaging in detection of gastric cancer precursors, as well as oesophageal and duodenal lesions.

DETAILED DESCRIPTION:
Gastric cancer is the fifth most common cause of death worldwide. Early detection and removal of gastric cancer precursors and early gastric cancer is crucial for good outcomes. However, these lesions are subtle and often missed by conventional white light imaging (WLI) endoscopy. Image enhanced endoscopy techniques have been developed to enhance the detection and characterization of gastrointestinal lesions. Narrow band imaging (NBI) is one such technique. Though widely used, its drawbacks include a limited far view as a result of the optical filter causing a dark endoscopic view. Linked color imaging (LCI) is a more recent image enhanced endoscopy technique that acquires images by using both narrow-band wavelength light and white light in an appropriate balance, enhancing slight color differences in the red region of mucosa. It has been proven to improve detection of H pylori gastritis and colorectal neoplasms. Thus far, there has been no study to determine whether the use of LCI will increase the detection rate of gastric cancer precursors and early gastric cancer compared to WLI. This study aims to determine whether LCI can increase the detection rate of gastric cancer precursors and early gastric cancer when compared to white light endoscopy, with the null hypothesis being no difference in detection rates. This study will also examine the use of LCI with magnification to predict histology findings for focal lesions seen on endoscopy, as well as the use of LCI in identifying esophageal lesions (such as Barett's esophagus) and duodenal lesions.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 50 years and above
* Patients undergoing gastroscopy for symptom evaluation
* Patients undergoing gastroscopy for surveillance of known intestinal metaplasia

Exclusion Criteria:

* Emergent gastroscopy performed for suspected acute GI bleeding
* Patients with previous surgical/endoscopic resection in stomach
* Patients with deranged coagulation and platelet function (INR>1.5, Plt<50)
* Patients with severe comorbid illness (ASA 3 and above)

Ages: 50 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2019-03-27 (Actual); Primary Completion 2020-10-17 (Actual); Study Completion 2020-10-17 (Actual)

PRIMARY OUTCOMES:
Difference in detection rate of gastric lesions between Linked Color Imaging and White Light Imaging | Immediately following the procedure
  Includes Intestinal Metaplasia, Gastric Adenoma, Low Grade Dysplasia, High Grade Dysplasia, Early Gastric Cancer
Difference in detection rate of oesophageal lesions between Linked Color Imaging and White Light Imaging | Immediately following the procedure
  Includes Barrett's Oesophagus, Low Grade Dysplasia, High Grade Dysplasia, Early Oesophageal Cancer
Difference in detection rate of duodenal lesions between Linked Color Imaging and White Light Imaging | Immediately following the procedure
  Includes Duodenal adenoma, Duodenal adenocarcinoma

SECONDARY OUTCOMES:
Sensitivity and Specificity of detection of gastric lesions | Upon histological confirmation - within 2 weeks of the procedure
  Includes Intestinal Metaplasia, Gastric Adenoma, Low Grade Dysplasia, High Grade Dysplasia, Early Gastric Cancer
Sensitivity and Specificity of detection of oesophageal lesions | Upon histological confirmation - within 2 weeks of the procedure
  Includes Barrett's Oesophagus, Low Grade Dysplasia, High Grade Dysplasia, Early Oesophageal Cancer
Sensitivity and Specificity of detection of duodenal lesions | Upon histological confirmation - within 2 weeks of the procedure
  Includes Duodenal adenoma, Duodenal adenocarcinoma

CONTACTS AND LOCATIONS:
Overall Officials: Tiing Leong Ang, MBBS, Principal Investigator — Changi General Hospital
Locations (2):
- Singapore (2):
  - Singapore General Hospital, Singapore
  - Changi General Hospital, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Dohi O, Yagi N, Onozawa Y, Kimura-Tsuchiya R, Majima A, Kitaichi T, Horii Y, Suzuki K, Tomie A, Okayama T, Yoshida N, Kamada K, Katada K, Uchiyama K, Ishikawa T, Takagi T, Handa O, Konishi H, Naito Y, Itoh Y. Linked color imaging improves endoscopic diagnosis of active Helicobacter pylori infection. Endosc Int Open. 2016 Jul;4(7):E800-5. doi: 10.1055/s-0042-109049. PMID 27556101
- [Result] Paggi S, Mogavero G, Amato A, Rondonotti E, Andrealli A, Imperiali G, Lenoci N, Mandelli G, Terreni N, Conforti FS, Conte D, Spinzi G, Radaelli F. Linked color imaging reduces the miss rate of neoplastic lesions in the right colon: a randomized tandem colonoscopy study. Endoscopy. 2018 Apr;50(4):396-402. doi: 10.1055/a-0580-7405. Epub 2018 Mar 14. PMID 29539651
- [Result] Yao K. The endoscopic diagnosis of early gastric cancer. Ann Gastroenterol. 2013;26(1):11-22. PMID 24714327
- [Result] Sun X, Dong T, Bi Y, Min M, Shen W, Xu Y, Liu Y. Linked color imaging application for improving the endoscopic diagnosis accuracy: a pilot study. Sci Rep. 2016 Sep 19;6:33473. doi: 10.1038/srep33473. PMID 27641243